CLINICAL TRIAL: NCT07029269
Title: Feasibility of Enhanced Recovery After Surgery Without Prophylactic Abdominal Drainage Tubes After Laparoscopic Distal Gastrectomy For Gastric Cancer: A Prospective, Multicenter, Non-inferiority, Randomized, Open-label, Controlled Trial
Brief Title: Feasibility of Enhanced Recovery After Surgery Without Prophylactic Abdominal Drainage Tubes After Laparoscopic Distal Gastrectomy For Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zuoyi Jiao (Other)
Responsible Party: Sponsor-Investigator, Zuoyi Jiao, Medical Professor, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LanzhouU2H-2025A-540
Record Dates: First submitted 2025-05-24; First posted 2025-06-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Gastric Adenocarcinoma; Laparoscopic Gastrectomy; Complications
Keywords: Enhanced Recovery After Surgery; tubeless; gastric adenocarcinoma; laparoscopic distal gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS-tubeless group (Experimental): Nasogastric decompression tube is not placed preoperatively; If necessary, nasogastric decompression tube is placed after anesthesia induction during surgery and removed when the reconstruction is performed; No abdominal drainage and nasojejunal feeding tubes were placed intraoperatively; None of these 3 tubes were present postoperatively.
  Interventions: Procedure: ERAS-tubeless group
- ERAS-tube group (Active Comparator): Nasogastric decompression tube is not placed preoperatively; If necessary, nasogastric decompression tube is placed after anesthesia induction during surgery and removed when the reconstruction is performed; Nasojejunal feeding tube is not placed intraoperatively; 1 prophylactic abdominal drainage tube is placed at the duodenal stump for LDG and retained postoperatively.
  Interventions: Procedure: ERAS-tube group

INTERVENTIONS:
Procedure: ERAS-tubeless group — Nasogastric decompression tube is not placed preoperatively; If necessary, nasogastric decompression tube is placed after anesthesia induction during surgery and removed when the reconstruction is performed; No abdominal drainage and nasojejunal feeding tubes were placed intraoperatively; None of these 3 tubes were present postoperatively.
  Arms: ERAS-tubeless group
Procedure: ERAS-tube group — Nasogastric decompression tube is not placed preoperatively; If necessary, nasogastric decompression tube is placed after anesthesia induction during surgery and removed when the reconstruction is performed; Nasojejunal feeding tube is not placed intraoperatively; 1 prophylactic abdominal drainage tube is placed at the duodenal stump for LDG and retained postoperatively.
  Arms: ERAS-tube group

SUMMARY:
This study aims to compare the effects of using prophylactic abdominal drainage tubes during Enhanced Recovery After Surgery (ERAS) in patients undergoing Laparoscopic Distal Gastrectomy (LDG) for gastric cancer through a multicenter non-inferiority randomized trial. The study is divided into two groups: 1. ERAS-tubeless group: The ERAS protocol without nasogastric decompression, nasojejunal feeding or prophylactic abdominal drainage tubes. 2. ERAS-tube group: the ERAS protocol with prophylactic abdominal drainage tubes, along with no nasogastric decompression or nasojejunal feeding tubes. Patients will be randomly assigned to the two groups in a 1:1 ratio, with the primary analysis based on the modified intention-to-treat population (mITT) and secondary analysis on the per-protocol (PP) population. Perioperative management will adhere to ERAS guidelines, and postoperative quality of life will be assessed using the EORTC QLQ-C30 questionnaire and QoR-15 scores. Preliminary training on the standard ERAS protocol is administered to all members in the team before the initiation of the study, ensuring in-group members to fully master the requirements and other related contents in the study. Data collectors, analysts, and outcome evaluators will remain blinded to group allocation. The findings of this study are expected to provide high-quality evidence on the feasibility of omitting prophylactic abdominal drainage in the context of ERAS, thereby contributing to the optimization of postoperative management strategies for gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age from 18 to 80 years old;
2. Histopathologically confirmed gastric adenocarcinoma;
3. Clinical tumor stage of cT1-4N0-3M0;
4. Laparoscopic distal gastrectomy approach;
5. ECOG score of 0-1;
6. Written informed consent

Exclusion Criteria:

1. Patients with severe concurrent illness or comorbid diseases;
2. Patients with severe pyloric obstruction, recurrent or remnant gastric cancer; 3. Patients with perforation, or undergoing emergency surgery;

4. Patients with a history of radiotherapy; 5. Patients undergoing complex abdominal surgeries other than laparoscopic cholecystectomy or appendectomy; 6. Patients with peritoneal, hepatic or ovarian metastasis, or simultaneous tumors in other parts of the body preoperatively and intraoperatively; 7. Patients with diabetes and poor recent glycemic control; 8. Patients with autoimmune diseases who have received corticosteroid treatment; 9. Patients with a BMI ≥30 kg/m2 or <18 kg/m2; 10. Patients with gastrointestinal hemorrhage and hemoglobin levels below 90 g/L; 11. Patients with hypoproteinemia and albumin levels below 30 g/L; 12. Patients with portal hypertension; 13. Patients with severe edema or dense fibrosis intraoperatively after neoadjuvant therapy; 14. Patients with intraoperative findings of duodenal invasion; 15. Patients with combined organ resection; 16. Reconstruction different from BillrothⅡand Braun anastomosis; 17. Patients with preoperative pathological examination inconsistent with postoperative result; 18. Declined to participate; 19. Patients with poor compliance and withdrew from the study halfway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 454 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of reoperation and/or percutaneous drainage placement by the 30th postoperative day. | The 30th day after surgery
  It refers to the total proportion of patients who, by the 30th day after their surgery, undergo either a reoperation or the placement of a percutaneous drainage device. The cumulative incidence considers all patients who experience one or both of these outcomes by the 30th day after surgery, providing insight into the postoperative recovery process.

SECONDARY OUTCOMES:
Postoperative hospital stay | It is expected to take 6 to 10 days
  Postoperative hospital stay is considered as a period from the time when a patient leaves the operating room to the point of time (8:00 am) on the day of discharge with no intervention treatment provided.
Overall 30 days morbidity or in hospital if longer than 30 days. | The 30th day after surgery
  The intraoperative complications include surgery-related complications (intraoperative hemorrhage (≥400 mL) and injury of liver, spleen, pancreas, and other vital organs), pneumoperitoneum-related complications (hypercapnia, mediastinal emphysema, subcutaneous emphysema, and respiratory and circulatory instability caused by pneumoperitonum), and anesthesia-related complications (acute bronchospasm, aspiration, abnormal blood pressure and temperature, and allergic reaction). The postoperative complications are defined as any adverse events requiring surgical or medical interventions after surgery, including surgery-related complications (wound problems, anastomotic leakage, anastomotic hemorrhage, anastomotic stenosis, intra-abdominal hemorrhage, intra-abdominal abscess, ileus, gastroparesis, lymphatic leakage, unscheduled reoperation, and surgery-related readmission) and system-related complications (pulmonary infection, pulmonary embolism, cardio-cerebrovascular complications (includ
30 days readmission rate and overall 90 days mortality. | Postoperative Day 30 and Day 90
  The 30 days readmission rate refers to the proportion of patients who are readmitted to a healthcare facility within 30 days after being discharged, attributable to postoperative complications. It is often used as a quality metric to assess healthcare effectiveness and the likelihood of complications or inadequate discharge planning. A higher readmission rate may indicate potential issues with the quality of care or patient management after discharge. The overall 90 days mortality refers to the proportion of patients who die within 90 days of either being admitted to or discharged from a healthcare facility, directly attributable to gastric cancer progression or surgery-related complications. This metric is used to evaluate the long-term survival rate of patients following their hospitalization and can serve as an indicator of the severity of the condition being treated, the effectiveness of treatment, and the overall healthcare system's ability to manage patients' long-term outcomes.
EORTC QLQ-C30 | Baseline, Postoperative Day 7 and Day 30
  EORTC QLQ-C30 questionnaire scale is used to assess the quality of life in both two groups. The assessment will be performed preoperatively (baseline), and at 7th day and 1 month after surgery.
Quality of postoperative recovery. | Baseline, Postoperative Day 1, Day 2, Day 3, Day 4, Day 5, and the Day of Discharge
  QoR-15 score is applied to evaluate the quality of recovery in both two groups. The evaluation will be conducted preoperatively (baseline), at 1st, 2nd, 3rd, 4th, 5th day after surgery and the day of discharge separately.
Time to first ambulation, time to first flatus, and time to first liquid diet. | It is expected to take 1 to 5 days.
  These time are defined as periods from the time when patients first return to the department after surgery to first out-of-bed activities, first anal exhaust, and first drinking sodium chloride aqueous solution separately. Operative time is defined as the interval from skin incision to skin closure.
NRS score. | The period is from the day of surgery to the day of discharge, which is expected to be approximately 7 days.
  Postoperative pain intensity is evaluated using the NRS score (0-10) and classified as no pain (0), mild pain (1-3), moderate pain (4-6), and severe pain (7-10). It is recorded from the day of surgery to the day of discharge.
PNI value. | The period is from the day of surgery to the day of discharge, which is expected to be approximately 7 days.
  The prognostic nutritional index (PNI) is an indicator, used to evaluate the nutritional status of patients and predict the risk of postoperative complications. It is calculated as peripheral blood lymphocyte count (109/L) × 5 + serum albumin value (g/L).
Medical cost. | The period is from the date of hospital admission to discharge, which is expected to take approximately 8 days.
  It is calculated as the total amount of medical expenses during the hospital stay for patients. The medical costs were strictly controlled in accordance with relevant regulations of the healthcare system, including the sum of all medically related expenses incurred during the patient's stay, such as bed charges, treatment fees, diagnostic and laboratory costs, medication, nursing, supplies, and other related expenses.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - International Hospital of Pecking University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center Gansu Hospital, Lanzhou, Gansu
  - Zhejiang Cancer Hospital, Zhejiang, Hangzhou
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Xi'an City

IPD SHARING:
Plan to Share IPD: No